CLINICAL TRIAL: NCT05261594
Title: Effects of Caffeine on Anxiety, Emotional Processing, Approach-avoidance Behavior, and Interoception in Panic Disorder - a Double Blind Randomized Controlled Study
Brief Title: Effects of Caffeine on Anxiety, Emotional Processing, Approach-avoidance Behavior, and Interoception in Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-06451
Record Dates: First submitted 2022-01-26; First posted 2022-03-02 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Panic Disorder; Healthy
MeSH Terms: conditions — Panic Disorder | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: The study entails two sessions and uses a crossover design. Participants will be randomized to start with either the caffeine condition or the placebo condition. Participants will complete the second session with the other condition (the condition not allocated to in session 1).
  The study includes two arms: (a) participants with Panic disorder (estimated n=50; actual n=30) and (b) healthy controls (estimated n=50; actual n=53). Both arms (Panic disorder and healthy controls) will complete both conditions (caffeine and placebo condition) in randomized order.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Panic disorder (Other): Participants will be randomized to start with either the caffeine condition or placebo condition. Participants will complete session 2 with the other condition (condition not allocated to in session 1).
  Interventions: Dietary Supplement: Caffeine; Drug: Placebo
- Healthy controls (Other): Participants will be randomized to start with either the caffeine condition or placebo condition. Participants will complete session 2 with the other condition (condition not allocated to in session 1).
  Interventions: Dietary Supplement: Caffeine; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — Caffeine capsule 150 mg, oral intake
Drug: Placebo — Placebo capsule, oral intake

SUMMARY:
The current study is a placebo-controlled, double-blind, randomized controlled study using a cross-over design, including participants with Panic disorder and healthy controls.

The study's primary aim is to investigate the effects of caffeine (vs placebo) on self-reported anxiety and its impact on emotional reactivity and goal-directed behavior in individuals with Panic disorder (vs healthy controls). Emotional reactivity will be measured with self-reported emotions and skin conductance responses. Caffeine-induced effects on goal-directed behavior will be assessed using an approach-avoidance conflict paradigm and an effort-allocation task. The occurrence of panic attacks and panic-related symptoms will also be measured. Furthermore, the link between a genotype of ADORA2A (rs5751876 T/T) previously associated with caffeine-induced anxiety, and the anxiogenic effects of caffeine will also be explored. In addition, caffeine-induced changes in attention to interoceptive stimuli (bodily sensation such as pulse and respiration) and anxiety elicited by attention to interoceptive stimuli will be explored. A secondary aim is to examine the potential caffeine-induced effects and the impact of genetic variation in healthy participants (caffeine vs placebo).

DETAILED DESCRIPTION:
Hypotheses

Self-reported anxiety during resting state

* Participants with Panic disorder will report higher resting-state levels of anxiety and negative emotions during the caffeine condition vs the placebo condition.
* Participants with Panic disorder will report higher resting-state levels of caffeine-induced (caffeine > placebo) anxiety and negative emotions compared to healthy subjects.

Panic attacks

* The occurrence of panic attacks and panic-related symptoms will be higher among participants with Panic disorder than in healthy controls in both conditions (caffeine and placebo).

Genetic variation

* Carriers of adenosine A2A receptor (i.e., ADORA2A) polymorphism (rs5751876 T/T) will report higher levels of caffeine-induced (caffeine >placebo) anxiety and negative emotions, in both individuals with Panic disorder and healthy participants.

Attention to interoceptive stimuli and associated anxiety

* Participants with Panic disorder will report higher levels of attention towards interoceptive stimuli in the caffeine condition (vs placebo).
* Participants with Panic disorder will report higher levels of self-reported anxiety associated with experiencing interoceptive stimuli during the caffeine condition (vs placebo).
* Participants with Panic disorder will report higher levels of self-reported attention to interoceptive stimuli and anxiety associated with experiencing interoceptive stimuli compared to healthy participants, both in general (placebo condition) and after caffeine intake (caffeine vs placebo).

Exploratory research questions

Analyses of emotional reactivity, the approach-avoidance conflict task, and the effort-allocation task will be exploratory without directed hypotheses, due to lack of previous research on the effects of caffeine in patients with Panic disorder on these tasks. We will also conduct exploratory analyses to explore if 150 mg of caffeine (vs placebo) affect self-reported levels of positive emotions in patients with Panic disorder and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Panic disorder group: Primary diagnosis of panic disorder.

Healthy control group: No current or history of psychiatric disorders.

All participants (Panic disorder and healthy): Weekly caffeine consumption ≤ 300 mg.

Exclusion Criteria:

History of severe psychiatric disorder (e.g. schizophrenia). Somatic or neurological conditions (e.g. hypertension and heart condition). Ongoing treatment with psychotropic medication or treatment with psychotropic medication which has been discontinued within 2 months. Other ongoing treatments that may confound the results. Current drug or alcohol abuse/dependency. Habitual nicotine use. Uncorrected visual or hearing impairment. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-03-19 (Actual)

PRIMARY OUTCOMES:
Self-reported anxiety | Session 1 (day 1)
  Anxiety will be assessed before capsule (caffeine/placebo) intake, 30 minutes after intake during rest, and after each task with self-reported ratings on a scale from 0-100 (0=no anxiety - 100=extreme anxiety).
Self-reported anxiety | Session 2 (minimum of 36 hours after Session 1 (day 1) maximum of 14 days after Session 1 (day 1))
  Anxiety will be assessed before capsule (caffeine/placebo) intake, 30 minutes after intake during rest, and after each task with self-reported ratings on a scale from 0-100 (0=no anxiety - 100=extreme anxiety).

SECONDARY OUTCOMES:
Self-reported emotions | Session 1 (day 1)
  Self-reported emotions (fear, bodily discomfort, negative feelings and positive feelings) will be assessed before capsule (caffeine/placebo) intake, 30 minutes after intake during rest, and after each task with self-reported ratings on a scale from 0-100 (0=none - 100=extreme).
Self-reported emotions | Session 2 (minimum of 36 hours after Session 1 (day 1) maximum of 14 days after Session 1 (day 1))
  Self-reported emotions (fear, bodily discomfort, negative feelings and positive feelings) will be assessed before capsule (caffeine/placebo) intake, 30 minutes after intake during rest, and after each task with self-reported ratings on a scale from 0-100 (0=none - 100=extreme).
Skin conductance responses (SCR) | Session 1 (day 1)
  SCR:s will be used to assess emotional reactivity at the physiological level to emotional stimuli vs neutral stimuli (faces).
Skin conductance responses (SCR) | Session 2 (minimum of 36 hours after Session 1 (day 1) maximum of 14 days after Session 1 (day 1))
  SCR:s will be used to assess emotional reactivity at the physiological level to emotional stimuli vs neutral stimuli (faces).
Approach-avoidance behavior | Session 1 (day 1)
  Approach-avoidance behavior will be assessed through an approach-avoidance incentive conflict task.
Approach-avoidance behavior | Session 2 (minimum of 36 hours after Session 1 (day 1) maximum of 14 days after Session 1 (day 1))
  Approach-avoidance behavior will be assessed through an approach-avoidance incentive conflict task.
Effort-allocation | Session 1 (day 1)
  Effort-allocation for rewards will be assessed using an effort-allocation task.
Effort-allocation | Session 2 (minimum of 36 hours after Session 1 (day 1) maximum of 14 days after Session 1 (day 1))
  Effort-allocation for rewards will be assessed using an effort-allocation task.
Occurrence of panic attack | Session 1 (day 1)
  The occurrence of a panic attacks will be assessed according to the Diagnostical Statistical Manual (DSM-5) criteria for panic attacks and will be coded dichotomous as "Present" or "Not present".
Occurrence of panic attack | Session 2 (minimum of 36 hours after Session 1 (day 1) maximum of 14 days after Session 1 (day 1))
  The occurrence of a panic attacks will be assessed according to the Diagnostical Statistical Manual (DSM-5) criteria for panic attacks and will be coded dichotomous as "Present" or "Not present".
Panic symptoms | Session 1 (day 1)
  Panic symptoms will be assessed by counting the number of DSM-5- panic attack symptoms reported by the participant.
Panic symptoms | Session 2 (minimum of 36 hours after Session 1 (day 1) maximum of 14 days after Session 1 (day 1))
  Panic symptoms will be assessed by counting the number of DSM-5- panic attack symptoms reported by the participant.
Attention to interoceptive stimuli | Session 1 (day 1)
  Attention to interoceptive stimuli will be assessed using self-reported ratings on a scale from 0-100 (0=no attention - 100= full attention). Interoceptive stimuli are defined as bodily sensation such as pulse and respiration.
Attention to interoceptive stimuli | Session 2 (minimum of 36 hours after Session 1 (day 1) maximum of 14 days after Session 1 (day 1))
  Attention to interoceptive stimuli will be assessed using self-reported ratings on a scale from 0-100 (0=no attention - 100= full attention). Interoceptive stimuli are defined as bodily sensation such as pulse and respiration.
Anxiety associated with attention to interoceptive stimuli | Session 1 (day 1)
  Self-reported ratings of anxiety associated with attention to interoceptive stimuli (bodily sensation such as pulse and respiration) will be assessed using self reported ratings on a scale from (0= no anxiety - 100 = extreme anxiety)
Anxiety associated with attention to interoceptive stimuli | Session 2 (minimum of 36 hours after Session 1 (day 1) maximum of 14 days after Session 1 (day 1))
  Self-reported ratings of anxiety associated with attention to interoceptive stimuli (bodily sensation such as pulse and respiration) will be assessed using self reported ratings on a scale from (0= no anxiety - 100 = extreme anxiety)

OTHER OUTCOMES:
Expectancy ratings | Session 1 (day 1)
  Participants will be asked to report if they believed that they received placebo or caffeine and how certain they are on a scale from 0-100%
Expectancy ratings | Session 2 (minimum of 36 hours after Session 1 (day 1) maximum of 14 days after Session 1 (day 1))
  Participants will be asked to report if they believed that they received placebo or caffeine and how certain they are on a scale from 0-100%
Panic Disorder Severity Scale (PDSS) | 1-7 days prior to session 1 (internet)
  PDSS is a self-reported questionnaire that assesses the severity of Panic disorder; range 0-28, higher scores indicating more severe symptoms
Body Sensations Questionnaire (BSQ) | 1-7 days prior to session 1 (via internet)
  BSQ assesses body sensations present during aversive situations; range 17-85, higher scores indicating higher levels of body sensations
Multidimensional Assessment of Interoceptive Awareness (MAIA-2) | 1-7 days prior to session 1 (via internet)
  MAIA-2 is an 8-scale state-trait questionnaire with 37 items to measure multiple dimensions of interoception by self-report. The score of each scale is the the average of the items on each scale. Higher mean scores indicate higher levels on of the measured dimensions (Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness,Self-Regulation, Body Listening, and Trust) on a scale from 0-5 (0=never- 5=always), respectively
Anxiety Sensitivity Index (ASI) | 1-7 days prior to session 1 (via internet)
  ASI assesses anxiety sensitivity; range 0-64, higher scores indicating higher anxiety sensitivity
Spielberger State-Trait Anxiety Inventory (STAI-T) | 1-7 days prior to session 1 (via internet)
  STAI-T is a self-rated questionnaire assessing trait anxiety; range 20-80, higher scores represent higher levels of trait anxiety
Caffeine Expectancy Questionnaire (CaffEQ) | 1-7 days prior to session 1 (via internet)
  CaffEQ is a self-rated questionnaire that assesses expected effect of caffeine intake.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Frick, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala university, Department of Medical Sciences, Psychiatry, Uppsala, Sweden